CLINICAL TRIAL: NCT07149285
Title: Effect of Mandala Practice on Menopausal Symptoms and Quality of Life
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emine Karacan (Other)
Responsible Party: Sponsor-Investigator, Emine Karacan, Assistant Professor, Gaziantep Islam Science and Technology University
Organization: Gaziantep Islam Science and Technology University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Protocol No:2025/523
Record Dates: First submitted 2025-07-03; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Menopause Symptom Management; Quality of Life; Menopausal Symptoms
Keywords: menopause; mandala painting; menopausal symptoms; quality of life; nursing

STUDY DESIGN:
Intervention Model Description: Intervention Group:
  The content of the study and the mandala application will be explained to women diagnosed with menopause, and after obtaining consent, a personal information form and scales regarding menopause symptoms and quality of life will be applied (Pre-test). Then, participants will be given a sample and blank mandala, 12 colored crayons and a follow-up form. The mandala application will be done for 20-30 minutes every day for 15 days, and will be monitored by phone every other day. At the end of the process, the scales will be re-applied (post-test) and the follow-up forms will be collected.
  Control Group:
  After the participants are informed about the study and their consent is obtained, the same scales will be applied (Pre-test). They will be interviewed again 15 days later and the scales will be filled out again (Post-test). Mandalas and pencils will be given to those who want them at the end of the study for ethical reasons.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know which group (experimental or control) they are included in or the effectiveness of the method applied to the experimental group. The researchers implementing the intervention will not be involved in the data analysis phase; data analysis will be conducted by independent researchers who are unaware of the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group: Women diagnosed with menopause will be invited to the study through face-to-face interviews at the outpatient clinic. Information will be provided about the study and the mandala application; women who agree to participate in the study will be asked to fill out an informed consent form, personal information form, menopause symptoms and menopause-specific quality of life assessment scales. Sample mandalas, blank mandalas, 12 different color crayons and a mandala application follow-up form will be distributed to the participants. The mandala application will be performed by the participants for 20-30 minutes every day for 15 days. In the interim periods (every other day), the application will be monitored by phone. At the end of the 15th day, the participants will be interviewed face-to-face again, the follow-up form will be collected and the menopause symptoms and quality of life scales will be re-administered.
  Interventions: Other: Mandala coloring
- The control group (No Intervention): The control group will be informed about the study in face-to-face interviews with women who applied to the outpatient clinic and were diagnosed with menopause, and women who agreed to participate in the study will be given an informed consent form, a personal information form, and menopause-specific quality of life and menopause symptom assessment scales and asked to fill them out. The women will be interviewed again 15 days later and given the menopause-specific quality of life and menopause symptom assessment scales again and asked to fill them out. In addition, the benefits of the mandala application will be explained to the women in order to eliminate the ethical dilemma, and coloring pencils with mandalas will be given to women who want to do the application. The women's routine care and treatments will continue during the data collection period.

INTERVENTIONS:
Other: Mandala coloring — Intervention Group:
  The content of the study and the mandala application will be explained to women diagnosed with menopause, and after obtaining consent, a personal information form and scales regarding menopause symptoms and quality of life will be applied. Participants will be given a sample and blank mandala, 12 colored crayons and a follow-up form. The mandala application will be done for 20-30 minutes every day for 15 days, and will be monitored by phone every other day. At the end of the process, the scales will be re-applied and the follow-up forms will be collected. Their routine treatments will continue.
  Arms: Intervention Group

SUMMARY:
Menopause is a natural cycle of life that mostly develops due to changes in the endocrine glands of the female body during middle age, and the menstrual cycle is permanently interrupted as a result of the ovaries losing their activity. Many symptoms are observed in women during menopause, and these symptoms cause women to experience many physiological, mental, social and sexual problems in the short or long term and to deteriorate their quality of life. In reducing the menopause symptoms experienced by women, hormone replacement therapy, traditional methods, mental or physical applications; aromatherapy, hypnosis, Biofeedback and relaxation techniques are used. The aim of these applications; is to relax women, reduce menopausal symptoms and increase their quality of life. Mandala, which has been widely used in the field of therapy in the past and today, is seen as a meditation tool in art therapy and is defined as a complementary, safe and accessible activity that supports mental health. It has been determined that how the mandala method, which is used in many areas in the literature, affects the symptoms and quality of life of women in the menopausal period has not been examined. For this reason, it is thought that this study will make a significant contribution to the literature.

DETAILED DESCRIPTION:
This study was designed as a randomized controlled experimental trial to examine the effects of mandala practice on menopausal symptoms and quality of life. The study will be conducted with 78 women (experimental = 39, control = 39) diagnosed with menopause at the Private Palmiye Hospital Gynecology and Obstetrics Outpatient Clinics. Participants will be randomly assigned to groups via random.org. Women in the experimental group will practice mandala coloring for 20-30 minutes daily for 15 days, while the control group will only be administered the scales and will be advised to practice mandala practice at the end of the study due to ethical principles. Data will be collected using a Personal Information Form, the Menopause Symptoms Assessment Scale, the Menopause-Specific Quality of Life Scale, and the Mandala Practice Follow-up Form. Data will be analyzed using frequency, descriptive statistics, the Shapiro-Wilks normality test, the independent samples t-test, one-way analysis of variance, and the Pearson correlation test in SPSS 24.0. It is anticipated that the findings of the study will make a significant contribution to the literature by revealing the effect of mandala practice in reducing symptoms and improving quality of life in menopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. The study included women who met the following conditions:
2. Absence of cognitive, hearing, or speech impairments that could interfere with effective communication,
3. No physical, psychological, or visual limitations that could hinder participation in mandala coloring activities,
4. Literacy in Turkish, including the ability to read, comprehend, and write,
5. A confirmed medical diagnosis of menopause,
6. Not undergoing any form of psychotherapy or alternative treatment throughout the study period,
7. Voluntary participation with signed informed consent.

Exclusion Criteria:

1. Participants were excluded from the study if they:
2. Provided incomplete or inaccurate responses in the data collection forms,
3. Were receiving hormone therapy to manage menopausal symptoms,
4. Had a neurological disorder that could impair concentration or communication during the mandala activity,
5. Had known allergies to paints or similar substances.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women diagnosed with menopause
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Menopausal Symptoms Assessment Scale (MSAS) total score | Pre-intervention (day 0) and post-intervention (day 15)
  Evaluation of the effect of mandala practice on the severity of somatic, psychological and urogenital symptoms in menopausal women. The MSAS consists of 11 items and three subscales. The subscales are labeled "Somatic Complaints," "Psychological Complaints," and "Urogenital Complaints." The scale is answered on a 5-point Likert-type scale, with each item scored as follows: 0: None, 1: Mild, 2: Moderate, 3: Severe, and 4: Extremely severe. The lowest possible score for the entire scale is 0, and the highest is 44. A higher total score indicates an increase in the severity of the complaints and a negative impact on quality of life.

SECONDARY OUTCOMES:
Menopause-Specific Quality of Life Scale (MSQL) total and sub-dimension scores | Pre-intervention (day 0) and post-intervention (day 15)
  Evaluation of the effect of mandala practice on the quality of life (vasomotor, psychosocial, physical and sexual dimensions) of menopausal women. The scale consists of four domains: vasomotor, psychosocial, physical, and sexual. It contains 29 Likert-type statements. As the score increases, the severity of the complaint and the quality of life decrease. Because the total scale uses an average score, the lowest possible score is 0, and the highest is 6. Each subdomain on the MSQL is scored from 0 to 6. A score of "0" indicates that no problem is experienced. A score of "1" indicates that the problem exists, but it is not bothersome at all. Scores between "2 and 6" indicate the severity and increasing severity of the problem.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Karacan, Asst Prof, Study Chair — Gaziantep Islamic Science and Technology University
Locations (1):
- Private Palmiye Hospital, Gynecology and Obstetrics Clinic, Hatay, İskenderun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not planned to share individual participant data collected in this study. This is because participant privacy was not protected and explicit consent for data sharing was not obtained. In addition, due to the sensitive nature of the data and ethical responsibilities, it was not deemed appropriate to share it with third parties.

REFERENCES:
- See also: Study Rationale and References — https://turkmedline.net/detay/menopoz-tutum-degerlendirme-olcegirsquonin-gecerlilik-ve-guvenilirlik-calismasi-eskisehir-mahmudiyersquode-40-64-yas-grubu-kadinlar-uzerinde-bir-calisma/76ba815200654b78/tr/342
- See also: Study Rationale and References — https://dergipark.org.tr/tr/pub/sdusbed/issue/44044/472704
- See also: Study Rationale and References — https://pubmed.ncbi.nlm.nih.gov/30868921/
- See also: Study Rationale and References — https://pubmed.ncbi.nlm.nih.gov/34403019/
- See also: Study Rationale and References — https://pubmed.ncbi.nlm.nih.gov/25932840/
- See also: Study Rationale and References — https://dergipark.org.tr/tr/pub/bpd/issue/60687/896437
- See also: Study Rationale and References — https://search.trdizin.gov.tr/tr/yayin/detay/384649/menopoz-semptomlarina-yoganin-etkisi?view=ris&download=384649.ris

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT07149285/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT07149285/ICF_001.pdf